CLINICAL TRIAL: NCT00308594
Title: Oral Dexamethasone for the Treatment of Cervical Radiculopathy: A Double Blinded, Randomized, Placebo Controlled Trial
Brief Title: Oral Dexamethasone for the Treatment of Cervical Radiculopathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to withdrawl of participating co-investigators.
Sponsor: University of Manitoba (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: B2006:027
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Cervical Radiculopathy
Keywords: cervical radiculopathy; dexamethasone; corticosteroid; oral
MeSH Terms: conditions — Radiculopathy | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dexamethasone

SUMMARY:
The purpose of this study is to determine whether dexamethasone is effective in the treatment of pain and disability resulting from a compressed spinal nerve in the neck (cervical radiculopathy).

DETAILED DESCRIPTION:
Cervical radiculopathy is causes both short and long term pain and diability. The current proven treatments include pain killers or surgery if there if patients experience progressive weakness or signs or spinal cord compression. Observations in both animal models and humans indicate that there is an inflammatory component to it. Corticosteroids (such as dexamethasone)are potent anti-inflammatories which may benefit people suffering from this condition. There is some evidence to support neck injections of drug directly onto the nerve root. This mmethod of drug delivery has been implicated with some serious complications such as paralysis and stroke. Delivering these medications in a pill form may provide a similar benefit without some of the serious complications.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 60
* arm and neck pain consistent with cervical radiculopathy
* Neck Disability Index score of at least 15 (moderate)
* symptom onset between 2 weeks and 6 months prior to enrollment

Exclusion Criteria:

* Actively immunosuppressed state
* clinical red flags consistent with possible infection or malignancy
* acute febrile illness or infection requiring antibiotics
* upper motor neuron signs consistent with myelopathy
* previous orthopedic neck surgery in the area of that nerve root
* known hepatic dysfunction
* schizophrenia
* pregnancy/nursing mothers
* previous chronic corticosteroid use
* diabetes mellitus on treatment
* rapidly improving course
* osteoporosis
* hypersensitivity to product components
* systemic fungal infection
* recent administration of live vaccine
* active tuberculosis
* glaucoma
* peptic ulcer disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index

SECONDARY OUTCOMES:
Visual Numeric Scale for arm & neck pain
Days missed from work
Cervical Radiculopathy Neurologic Impairment Scale

CONTACTS AND LOCATIONS:
Overall Officials: Dave R Hooper, MD BSc, Principal Investigator — University of Manitoba